CLINICAL TRIAL: NCT07384572
Title: Evaluation of Perioperative Recovery Outcomes of a Spontaneous Breathing-Preserving Strategy in Severely Underweight Lung Transplantation: A Prospective, Multicenter, Single-Arm Clinical Study
Brief Title: Perioperative Recovery Outcomes With a Spontaneous Breathing Strategy in Severely Underweight Lung Transplant Recipients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Chief Physician and Professor of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BREATHE-LowWt
Record Dates: First submitted 2026-01-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: End-stage Lung Disease
Keywords: Lung transplantation; Enhanced Recovery After Surgery; Severely Underweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tubeless LTx Group (Experimental): All participants receive lung transplantation under a standardized spontaneous-breathing-preserving ("tubeless") pathway. After anesthesia induction, a supraglottic airway (laryngeal mask airway) is used when feasible with regional nerve blocks and multimodal sedation/analgesia to control pain and cough while maintaining spontaneous breathing. Muscle relaxants are minimized; ventilatory assistance is provided only as needed with low airway pressures. Postoperatively, patients are managed in the intensive care unit with spontaneous breathing and protocol-guided noninvasive respiratory support. Conversion to endotracheal intubation, invasive mechanical ventilation, and/or extracorporeal membrane oxygenation is allowed if predefined safety criteria are met.
  Interventions: Procedure: Lung transplantation that preserves spontaneous breathing function

INTERVENTIONS:
Procedure: Lung transplantation that preserves spontaneous breathing function — This intervention uses a spontaneous-breathing-preserving anesthesia strategy during lung transplantation, which differs from conventional management based on endotracheal intubation and invasive mechanical ventilation. A supraglottic airway (laryngeal mask airway) is used when feasible instead of endotracheal intubation to maintain spontaneous breathing throughout the procedure. Neuromuscular blocking agents are minimized, and regional nerve blocks (such as intercostal nerve blocks or paravertebral blocks) are used to control pain and suppress cough while preserving the patient's ability to breathe independently. After surgery, patients receive protocol-guided noninvasive respiratory support (for example, high-flow nasal oxygen or noninvasive ventilation), with the goal of avoiding routine invasive mechanical ventilation.

SUMMARY:
The goal of this prospective, multicenter, single-arm clinical study is to learn whether a spontaneous breathing-preserving perioperative management strategy can improve recovery and is safe in lung transplant recipients with very low body weight (body mass index [BMI] <16 kg/m²).

The main questions it aims to answer are whether, in lung transplant recipients with very low body weight (BMI <16 kg/m²), a spontaneous breathing-preserving anesthesia-surgical strategy combined with standardized nutritional optimization and a prehabilitation program can improve early postoperative recovery and perioperative survival. Specifically, the study will assess the proportion of participants who require postoperative invasive mechanical ventilation, postoperative length of hospital stay, and perioperative survival within the protocol-defined time window (e.g., through hospital discharge).

Participants will undergo lung transplantation using a perioperative strategy that preserves spontaneous breathing whenever clinically appropriate, with predefined criteria for conversion to endotracheal intubation and mechanical ventilation if needed. They will receive standard postoperative monitoring and supportive care, with respiratory support events and perioperative complications assessed during the index hospitalization (and up to 30 days after surgery, if specified in the protocol). Key outcomes will be collected from routine clinical care, including postoperative ventilatory support status, length of hospital stay, and major safety events.

DETAILED DESCRIPTION:
This prospective, multicenter, single-arm clinical study will evaluate the clinical effectiveness and safety of a spontaneous breathing-preserving anesthesia-surgical strategy, integrated with standardized nutritional optimization and a structured prehabilitation program, in lung transplant recipients with very low body weight (body mass index [BMI] <16 kg/m²). The overall purpose is to determine whether this bundled perioperative approach can enhance early postoperative recovery while maintaining acceptable perioperative survival in this high-risk population.

Eligible participants will be enrolled consecutively across participating centers and managed according to a standardized perioperative pathway. The intervention bundle includes: (1) preoperative nutritional optimization and prehabilitation tailored to severe low BMI status, and (2) an intraoperative anesthesia-surgical management strategy designed to preserve spontaneous breathing whenever clinically appropriate, with predefined criteria for escalation/conversion to endotracheal intubation and invasive mechanical ventilation (IMV) if safety thresholds are exceeded. Postoperatively, participants will receive standard monitoring and supportive care per institutional lung transplant practice, with protocolized collection of key respiratory support events and perioperative complications. Outcomes will be assessed during the index hospitalization and, where specified by the protocol, through a defined perioperative follow-up window (e.g., up to 30 days after surgery).

The primary clinical outcomes focus on early recovery and perioperative survival: (1) the proportion of participants requiring postoperative IMV, (2) postoperative length of hospital stay, and (3) perioperative survival within the protocol-defined time window (e.g., through hospital discharge and/or up to 30 days). Additional safety and recovery measures may include intensive care unit length of stay, re-intubation or tracheostomy, new or escalated extracorporeal support, primary graft dysfunction grading at prespecified time points, infections, airway complications, bleeding requiring re-intervention, acute kidney injury and renal replacement therapy, major cardiovascular/cerebrovascular events, and rejection episodes. Analyses will primarily be descriptive and estimation-focused, reporting event rates, central tendencies for length-of-stay outcomes, and survival estimates with confidence intervals; where appropriate, findings may be contextualized against prespecified benchmarks or contemporaneous historical outcomes.

The study is expected to generate high-quality prospective evidence on the feasibility and clinical signals of benefit of a spontaneous breathing-preserving perioperative strategy in severely underweight lung transplant recipients. It is hypothesized that the bundled approach will be associated with a lower need for postoperative IMV and shorter postoperative hospitalization, while maintaining acceptable perioperative survival and safety profiles in this vulnerable population. Results are intended to inform standardized perioperative pathways and support broader implementation and future comparative studies.

ELIGIBILITY:
[1] Inclusion Criteria

1. Age and informed consent: Age ≥18 years; able to understand the study and provide written informed consent; willing and able to comply with follow-up.
2. Transplant candidacy: Listed in CLuTR or the participating center's lung transplant waiting list and scheduled to undergo allogeneic lung transplantation.
3. Low body weight definition (core cohort criterion): Preoperative BMI <16 kg/m², calculated using the most recent traceable preoperative height and weight within the evaluation window.
4. Preoperative support status: Not receiving ongoing invasive mechanical ventilation (endotracheal intubation or tracheostomy) and not on ECMO or other extracorporeal life support preoperatively.
5. Minimum acceptable end-organ function: LVEF ≥40%; eGFR ≥40 mL/min/1.73 m²; no evidence of acute liver failure or decompensated cirrhosis/portal hypertension; American Society of Anesthesiologists (ASA) physical status ≤ IV.
6. Infection and transmissible diseases: No evidence of active infection; no active tuberculosis; HIV/HBV/HCV status meeting center transplant requirements (e.g., undetectable viral load, where applicable).
7. Rehabilitation and support: Demonstrated potential for postoperative rehabilitation (able to participate in training) and reliable caregiving support (at least one primary caregiver).

[2] Exclusion Criteria

1. Consent/compliance: Refusal or withdrawal of informed consent; investigator judgment that follow-up cannot be completed or presence of recurrent severe non-adherence.
2. Transplant type: Retransplantation, multi-organ transplantation, or planned lobar lung transplantation.
3. Recent major cardiovascular/cerebrovascular events: Acute coronary syndrome/myocardial infarction or stroke within the past 30 days.
4. Severe organ dysfunction/acute failure: LVEF <40%; eGFR <40 mL/min/1.73 m²; acute liver failure or decompensated cirrhosis/portal hypertension; acute renal failure requiring dialysis with low likelihood of recovery; significant preoperative neuropsychiatric disorder or altered mental status.
5. High-risk/severe infection: Septic shock; active extrapulmonary or disseminated infection; active tuberculosis; detectable HIV viral load (or otherwise not meeting center transplant standards).
6. High bleeding risk: Severe bronchiectasis not treated with preoperative vascular intervention or not readily correctable.
7. Malignancy: Active malignancy or malignancy with high risk of recurrence or cancer-related mortality.
8. Severe chest wall or spinal deformity: Definitively diagnosed severe thoracic cage deformity or spinal deformity.
9. Substance use/dependence: Current use of cigarettes, e-cigarettes, inhaled cannabis, or intravenous drugs.
10. Tubeless/spontaneous breathing-preserving strategy not safely feasible: Determined by the anesthesia team to have a difficult airway or unsafe supraglottic/non-intubated airway management (e.g., anticipated intraoperative airway difficulty, pharyngeal/laryngeal narrowing not suitable for a laryngeal mask airway), including but not limited to: Mallampati class >III, mouth opening <3 cm, thyromental distance <5 cm, or significant airway anatomic variants (e.g., aberrant right upper lobe bronchial takeoff in a planned right lung transplant) deemed difficult to manage safely with an LMA or single-lumen tube.
11. Donor/donor lung limitations: Donor age >60 years; donor mechanical ventilation >14 days; positive donor airway microbiology deemed unacceptable by the transplant team.
12. Protected populations: Pregnant or breastfeeding women.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Requiring Postoperative Invasive Mechanical Ventilation (IMV) During Index Hospitalization | From ICU admission immediately after leaving the operating room until hospital discharge or in-hospital death, assessed up to 90 days postoperatively (if hospitalization extends beyond 90 days, events after day 90 will not be counted for this outcome).
  Number of participants who require postoperative invasive mechanical ventilation (IMV) delivered via an endotracheal tube or tracheostomy tube at any time after leaving the operating room and before hospital discharge (or in-hospital death).
Postoperative Hospital Length of Stay (Days) During Index Hospitalization | From end of surgery (postoperative Day 0) until hospital discharge or in-hospital death (index hospitalization), assessed up to 90 days.
  The number of days from the end of surgery (postoperative Day 0) to the date the participant is discharged from the index hospitalization, according to institutional discharge criteria. Participants who die in hospital will be assigned length of stay through the date of in-hospital death.
Rate of Perioperative Survival | From start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first.
  Perioperative survival is defined as the proportion of participants who remain alive from the start of transplant surgery through hospital discharge or postoperative Day 30, whichever occurs first. Participants who die before discharge or before postoperative Day 30 will be counted as non-survivors for this outcome.

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data (IPD) underlying the analyses of this clinical study, limited to baseline and perioperative variables. Baseline IPD will include demographics (e.g., age, sex), primary diagnosis, key comorbidities, and transplant-relevant preoperative measures and donor/recipient characteristics recorded in structured fields. Perioperative IPD will include operative and anesthesia strategy, airway management, intraoperative/early postoperative respiratory and hemodynamic parameters, major perioperative interventions (e.g., ECMO use), and key in-hospital outcomes during the index hospitalization (e.g., need for postoperative IMV, complications, ICU/hospital length of stay, and in-hospital mortality). The study protocol and statistical analysis plan will also be shared. All direct identifiers will be removed and dates will be shifted/aggregated as needed to protect privacy.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning at study completion and ending 2 years after study completion.
Access Criteria: De-identified IPD and supporting documents (study protocol, statistical analysis plan, and data dictionary) will be available to qualified researchers outside the primary study group for scientifically sound research purposes. Access will be granted upon submission of a written request that includes a brief research proposal, analysis plan, and proof of relevant ethics/IRB review if applicable. Requests will be reviewed by the study steering committee/data access committee. Approved requestors must sign a data use agreement prohibiting re-identification attempts and onward sharing, and requiring appropriate data security measures and acknowledgement of the original study. Data will be provided through a secure electronic transfer or a controlled-access online repository; access instructions will be provided after approval.
URL: https://www.gyfyyy.cn/